CLINICAL TRIAL: NCT03208179
Title: IPTp With Dihydroartemisinin-piperaquine and Azithromycin for Malaria, Sexually Transmitted and Reproductive Tract Infections in Pregnancy in High Sulphadoxine-pyrimethamine Resistance Areas in Kenya, Malawi and Tanzania
Brief Title: Improving PRegnancy Outcomes With Intermittent preVEntive Treatment in Africa
Acronym: IMPROVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Kenya Medical Research Institute (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); National Institute for Medical Research, Tanzania (Other Government); Kilimanjaro Christian Medical Centre, Tanzania (Other); University of Copenhagen (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); London School of Hygiene and Tropical Medicine (Other); University College, London (Other); Tampere University (Other); University of Bergen (Other); University of Massachusetts, Worcester (Other); University of Toronto (Other); University of Melbourne (Other); Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16.049
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy; Malaria in Pregnancy; Malaria
Keywords: Malaria in Pregnancy; Intermittent Preventive Treatment; IPTp
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be a partially placebo-controlled involving a single placebo for AZ. To further minimise bias, an objective primary outcome measure will be used and all staff will be masked to the treatment assignment of individual women. The trial statistician will also be masked in regard to the treatment code when he develops the statistical analysis plan and writes the statistical programmes, which will be validated and completed using dummy randomisation codes. The actual allocation will only be provided to the study team after locking of the database and approval of the statistical analysis plan by the independent Data Monitoring and Ethics Committee (DMEC) before they review any trial results. The study statistician conducting the interim analysis will remain masked throughout the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPTp-SP (Active Comparator): Stat course of 3 tablets of quality-assured SP (tablets of 500 mg of sulphadoxine and 25 mg of pyrimethamine) at each scheduled antenatal visit
  Interventions: Drug: sulphadoxine-pyrimethamine
- IPTp-DP (Experimental): Dihydroartemisinin-piperaquine [3 to 5 tablets of DP (tablets of 40 mg of dihydroartemisinin and 320 mg of piperaquine, based on bodyweight) daily for 3 days] + placebo AZ at each scheduled antenatal visit
  Interventions: Drug: dihydroartemisinin-piperaquine
- IPTp-DPAZ (Experimental): Dihydroartemisinin-piperaquine [3 to 5 tablets of DP (tablets of 40 mg of dihydroartemisinin and 320 mg of piperaquine, based on bodyweight) daily for 3 days] + AZ tablet [1.5g over 3 days as 500mg per day] at each scheduled antenatal visit.
  Interventions: Drug: dihydroartemisinin-piperaquine plus azithromycin

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — Women randomised to this intervention will receive 3 day treatment dose of dihydroartemisinin-piperaquine by body weight plus azithromycin placebo
  Other Names: Eurartesim
  Arms: IPTp-DP
Drug: sulphadoxine-pyrimethamine — Women randomised to this intervention will receive stat dose of 3 tablets of 500 mg sulphadoxine and 25 mg of pyrimethamine each (total dose of 1,500mg sulphadoxine and 75mg pyrimethamine) on a single day of clinic visit
  Other Names: Fansidar
  Arms: IPTp-SP
Drug: dihydroartemisinin-piperaquine plus azithromycin — Women randomised to this intervention will receive 3 day treatment dose of dihydroartemisinin-piperaquine by body weight plus azithromycin (500mg)
  Other Names: Eurartesim plus Zithromax
  Arms: IPTp-DPAZ

SUMMARY:
This study evaluates the efficacy and safety of monthly intermittent preventive treatment using dihydroartemisinin piperaquine (DP) alone or in combination with azithromycin (AZ) compared to sulphadoxine-pyrimethamine (SP) for the prevention of malaria in pregnant women in the second and third trimester.

DETAILED DESCRIPTION:
Intermittent preventive treatment with sulphadoxine-pyrimethamine (IPTp-SP) is one of the pillars of malaria prevention in pregnancy in sub-Saharan Africa, in addition to prompt case management and use of long lasting insecticide treated bednets. However, mounting resistance to SP by Plasmodium falciparum increasing renders IPTP-SP ineffective.

Two exploratory trials in Uganda and Kenya demonstrated that IPTp with DP was superior to IPTp-SP for the prevention of malaria infection in pregnancy. However, neither study was adequately powered to look at adverse birth outcomes. This study is a confirmatory efficacy trial in Malawi, Tanzania and Kenya to determine the efficacy and safety of IPTp with DP alone or in combination with AZ.

This will be a 3-arm trial, superiority, partial blinded, placebo controlled, randomized trial comparing IPTp with SP, versus IPTp with DP alone, and IPTp with DP+AZ with the following hypotheses:

* IPTp with DP is superior to IPTp with SP in preventing adverse pregnancy outcomes.
* The combination of DP with AZ further reduces adverse pregnancy outcomes compared to IPTp with DP alone.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 16-28 weeks' gestation
* Viable singleton pregnancy
* Resident of the study area
* Willing to adhere to scheduled and unscheduled study visit procedures
* Willing to deliver in a study clinic or hospital
* Provide written informed consent

Exclusion Criteria:

* Multiple pregnancies (i.e. twin/triplets)
* HIV-positive
* Known heart ailment
* Severe malformations or non-viable pregnancy if observed by ultrasound
* History of receiving IPTp-SP during this current pregnancy
* Unable to give consent
* Known allergy or contraindication to any of the study drugs

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant female
Enrollment: 4680 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | 8 months
  Composite of foetal loss (spontaneous abortion or stillbirth), or singleton live births born small-for-gestational age (SGA), or with low birthweight (LBW), or preterm (PT) (SGA-LBW-PT), or subsequent neonatal death by day 28.

SECONDARY OUTCOMES:
Composite of foetal loss and neonatal mortality | 8 months
  Composite of foetal loss (spontaneous abortion or stillbirth) and neonatal mortality
SGA-LBW-PT composite | 6 months
  Composite of small for gestational age, low birth weight or preterm birth
SGA | 6 months
  Small for gestational age using the new INTERGROWTH population reference's 10th percentile
LBW | 6 months
  Low birth weight defined as a corrected birth weight below 2.5 kg
PT | 6 months
  Preterm birth defined as birth at a gestational age above 28 weeks but less than 37 completed weeks
Neonatal length and stunting | 8 months
  Neonatal length and stunting
Clinical malaria during pregnancy | 6 months from randomisation
  Incidence of clinical malaria during pregnancy
Malaria infection during pregnancy detected by microscopy and PCR | 6 months from randomisation
  Prevalence and incidence of peripheral maternal (blood) malaria infection during pregnancy by microscopy and PCR
Composite placental malaria detected by microscopy, by molecular methods or by histology | 6 months from randomisation
  Prevalence of placental malaria by microscopy, PCR and placental histology
Placental malaria detected by microscopy | 6 months from randomisation
  Prevalence of placental malaria detected in maternal placental blood by microscopy
Placental malaria detected by molecular methods (PCR) | 6 months from randomisation
  Prevalence of placental malaria detected in maternal placental blood by PCR
Placental malaria detected by histology | 6 months from randomisation
  Prevalence of placental malaria detected in full placental section by histology
Maternal nutritional status | 6 months from randomisation
  Changes in maternal nutritional status by MUAC and BMI.
Maternal anaemia during pregnancy and delivery | 6 months from randomisation
  Prevalence and incidence of maternal anaemia (Hb < 11g/dl) at enrolment, last antenatal visit and delivery
Congenital anaemia | 6 months from randomisation
  Prevalence of anaemia (Hb < 13g/dl) from newborn cord blood
Congenital malaria infection | 6 months from randomisation
  Prevalence of malaria infection by microscopy or PCR from newborn cord blood
QTc-prolongation | 6 months from randomisation
  QTcF-prolongation of more than 60ms between baseline DTcF prior to first dose of DP (+/- AZ) on day 0 and repeat QTcF 4 - 6 hrs after administration of 3rd dose of DP(+/- AZ) on day 2, or QTcF > 480ms, 4 - 6 hours after on day 2 treatment administration. Only on the DP containing arms.
Congenital malformations | 6 months from randomisation
  Any visible external congenital abnormality on surface examination
Maternal mortality | 8 months from randomisation
  The death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes.
Other SAEs and AEs | 8 months from randomisation
  Incidence of AEs and SAEs
(History of) vomiting study drug | 6 months from randomisation
  Prevalence and incidence of vomiting investigational product (IP) twice at the same IP administration visit
Dizziness | 6 months from randomisation
  Prevalence of dizziness after a course of IP
Gastrointestinal complaints | 6 months from randomisation
  Prevalence of gastrointestinal complaints after a course of IP
Molecular markers of drug resistance in Plasmodium falciparum infections during pregnancy and delivery | 6 months from randomisation
  Prevalence and incidence of SP and artemisinin resistance markers from infection isolates after enrollment and at delivery
Presence of STIs/RTIs prior to delivery (syphilis, gonorrhoea, Chlamydia trachomatis, Trichomonas vaginalis, and bacterial vaginosis) | 6 months from randomisation
  Prevalence and incidence of STIs/RTIs (syphilis, gonorrhoea, Chlamydia trachomatis, Trichomonas vaginalis, and bacterial vaginosis) at randomization and last antenatal visit prior to delivery
Changes in macrolide resistance in Pneumococcus detected in maternal nasopharyngeal samples | 6 months from randomisation
  Prevalence and incidence of carriage of macrolide resistant pneumococcus at randomization and delivery
Changes in the colony composition of maternal vaginal microbiota, and intestinal microbiota of mother and infant. | 6 months from randomisation
  Changes in maternal reproductive tract and gut microbiota from randomisation to last antenatal visit prior to delivery, and neonatal gut microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Simon K Kariuki, PhD, Principal Investigator — Kenya Medical Research Institute; Frank Mosha, PhD, Principal Investigator — Kilimanjaro Christian Medical University College; John Lusingu, PhD, Principal Investigator — National Institute for Medical Research
Locations (7):
- Kenya (3):
  - Ahero Sud-countyHospital, Ahero, Kisumu County
  - Homa Bay County Hospital, Homa Bay
  - Rabour Sub-county Hospital, Kisumu
- Malawi (2):
  - Chikwawa District Hospital, Chikwawa
  - Mangochi District Hospital, Mangochi
- Tanzania (2):
  - Handeni District Hospital, Handeni
  - Korogwe District Hospital, Korogwe

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified participant data will be made available for meta-analyses as soon as the data analysis is completed, with the understanding that results of the meta-analysis will not be published prior to the results of the individual trial without prior agreement of the investigators. No later than 5 years after the publication of the trial a fully de-identified data set will be available for sharing purposes
Supporting Information: Study Protocol, ICF
Time Frame: No later than 5 years after publication
Access Criteria: Open access

REFERENCES:
- [Derived] Gore-Langton GR, Madanitsa M, Barsosio HC, Minja DTR, Mosha J, Kavishe RA, Mtove G, Gesase S, Msemo OA, Kariuki S, Otieno K, Phiri KS, Lusingu JPA, Mukerebe C, Manjurano A, Ikigo P, Saidi Q, Onyango ED, Schmiegelow C, Dodd J, Hill J, Hansson H, Alifrangis M, Gutman J, Hunter PJ, Klein N, Ashorn U, Khalil A, Cairns M, Ter Kuile FO, Chico RM. Prevalence and risk factors of curable sexually transmitted and reproductive tract infections and malaria co-infection among pregnant women at antenatal care booking in Kenya, Malawi and Tanzania: a cross-sectional study of randomised controlled trial data. BMJ Public Health. 2024 Sep 18;2(2):e000501. doi: 10.1136/bmjph-2023-000501. eCollection 2024 Dec. PMID 40018559
- [Derived] Madanitsa M, Barsosio HC, Minja DTR, Mtove G, Kavishe RA, Dodd J, Saidi Q, Onyango ED, Otieno K, Wang D, Ashorn U, Hill J, Mukerebe C, Gesase S, Msemo OA, Mwapasa V, Phiri KS, Maleta K, Klein N, Magnussen P, Lusingu JPA, Kariuki S, Mosha JF, Alifrangis M, Hansson H, Schmiegelow C, Gutman JR, Chico RM, Ter Kuile FO. Effect of monthly intermittent preventive treatment with dihydroartemisinin-piperaquine with and without azithromycin versus monthly sulfadoxine-pyrimethamine on adverse pregnancy outcomes in Africa: a double-blind randomised, partly placebo-controlled trial. Lancet. 2023 Mar 25;401(10381):1020-1036. doi: 10.1016/S0140-6736(22)02535-1. Epub 2023 Mar 10. PMID 36913959
- [Derived] Mtove G, Abdul O, Kullberg F, Gesase S, Scheike T, Andersen FM, Madanitsa M, Ter Kuile FO, Alifrangis M, Lusingu JPA, Minja DTR, Schmiegelow C. Weight change during the first week of life and a new method for retrospective prediction of birthweight among exclusively breastfed newborns. Acta Obstet Gynecol Scand. 2022 Mar;101(3):293-302. doi: 10.1111/aogs.14323. Epub 2022 Feb 13. PMID 35156190